CLINICAL TRIAL: NCT02863692
Title: Registry of the German CLL Study Group Long Term Follow-up of Patients With CLL, B-PLL, T-PLL, SLL,T or NK-LGL, HCL and Richter's Transformation
Brief Title: Registry of the German CLL Study Group
Acronym: CLL-Registry
Status: Recruiting | Type: Observational
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Other Study IDs: CLL-Registry
Record Dates: First submitted 2015-02-26; First posted 2016-08-11 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: CLL; SLL; HCL; Richter´s Transformation; Leukemia, Prolymphocytic, B-Cell; Leukemia, Prolymphocytic, T-Cell; T-LGL Leukemia; NK-LGL Leukemia
Keywords: CLL; B-PLL; T-PLL; SLL; T-NK-LGL; HCL; Richter´s Transformation
MeSH Terms: conditions — Leukemia, Prolymphocytic, B-Cell; Leukemia, Prolymphocytic, T-Cell; Leukemia, Large Granular Lymphocytic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Long term follow-up of patients with chronic lymphocytic leukemia (CLL), B-prolymphocytic leukemia (B-PLL), T-cell prolymphocytic leukemia (T-PLL), Small lymphocytic lymphoma (SLL), T/Natural Killer large granular lymphocyte leukemia (T or NK-LGL), Hairy cell leukemia (HCL) and Richter's transformation

DETAILED DESCRIPTION:
The most frequent primary endpoint in phase III trials of CLL is progression-free survival (PFS). However, the most important endpoint is overall survival (OS) which is usually a secondary endpoint in such trials. The outcome after progression is critical and responses to second and subsequent therapies may differ between the trial arms. Therefore it is essential to assess OS in addition to PFS. In addition, late toxicities, such as myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML), Epstein-Barr virus (EBV)-associated lymphoproliferative disease or Hodgkin's disease, late opportunistic infections and second malignancies, are increasingly seen and are likely to differ depending on the intensity of therapy. Moreover, meta-analysis of several phase III trials with long follow-periods are desirable. Similarly, valid analyses of biological disease characteristics in relation to outcome are depending on large collections of clinical data with mature follow-up.

The findings of the CLL8 study provide evidence that the addition of rituximab to chemotherapy with Fludarabine and Cyclophosphamide (FC) may prolong survival of patients with CLL. However, it also opens the question about whether applying such therapy might cause certain late toxicities and whether it improves longterm survival for patients with CLL. Moreover the outcome of subsequent therapies after various first line treatments with Fludarabine (F), FC, Bendamustine and Rituximab (BR) or Fludarabine, Cyclophosphamide and Rituximab (FCR) amongst others outside of clinical trials needs to be investigated further.

Recently published phase III trials in CLL showed median observation times ranging from 22 to 41 months, but most of the trials report observation times around 2 years only. For most of the phase III trials of the German CLL Study Group (GCLLSG) great efforts were made to implement an extended follow up in these trials, but due to administrative reasons the follow up is limited to at most 8 years. This registry should enable the collection of data of the entire course of diseases in- and outside of clinical trials.

Besides CLL other related rare lymphoproliferative malignancies will be included in this registry. On the one hand for historical on the other hand for clinical reasons these diseases are close to CLL and information about them should be gathered as best as possible.

Only limited information is available for patients with SLL, B-PLL, T-PLL, T/NK-LGL, HCL and Richter's transformation. They carry orphan disease status and long-term follow-up data is urgently needed.

To our knowledge there are no comparable registries for patients with CLL, B-PLL, T-PLL, SLL, T/NK-LGL, HCL or Richter's transformation. In order to understand and gain greater insight into the biology, the response to treatment and the outcome of very rare diseases it is extremely important to gather structured information about the patients and their disease centrally.

ELIGIBILITY:
Inclusion Criteria (all must apply)

1. Confirmed diagnosis of CLL, B-PLL, T-PLL, SLL, T or NK-LGL, HCL or Richter's transformation
2. 18 years of age or older
3. Signed, written informed consent
4. Presence of one or more of the following disease situations:

   * Newly diagnosed patients without treatment indication (eligible for watch and wait Approach Treatment within a clinical trial according to the AMG or status post participation in a clinical Trial)
   * Treatment with standard therapies approved for the eligible entities or status post treatment (outside of clinical trials)
   * Referral for evaluation the indication for HSCT
   * Relapsed disease status (even if first diagnosis was prior to activation of the registry)

Exclusion Criteria

1. Patients without confirmed diagnosis of CLL, B-PLL, T-PLL, SLL, T or NK- LGL, HCL or Richter's transformation
2. Cerebral dysfunction, legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of CLL, B-PLL, T-PLL, SLL, T or NK-LGL, HCL or Richter's transformation
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2013-08; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | from date of registry entry until date of death, up to 12 years
  Overall survival will be measured from date of registry entry until date of death

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Study Director — German CLL Study Group, Department I of Internal Medicine University Hospital Cologne
Locations (1):
- BAG Freiberg-Richter, Jacobasch, Wolf, Illmer, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kutsch N, Giza A, Robrecht S, Stumpf J, Federhen A, Stoltefuss A, Vehling-Kaiser U, Koenigsmann M, Tausch E, Schneider C, Stilgenbauer S, Illmer T, Schlag R, Dorfel S, Gaska T, Kiehl M, Muller-Hagen S, Moorahrend E, Linde H, Schlenska-Lange A, von Tresckow J, Fischer K, Eichhorst B, Hallek M, Fink AM. Fludarabine, cyclophosphamide, and rituximab as first-line treatment in patients with chronic lymphocytic leukemia: A long-term analysis of the German CLL Study Group (GCLLSG) registry. Eur J Haematol. 2024 Aug;113(2):235-241. doi: 10.1111/ejh.14220. Epub 2024 May 1. PMID 38693677
- [Background] Furstenau M, Giza A, Stumpf T, Robrecht S, Maurer C, Linde H, Jacobasch L, Dorfel S, Aldaoud A, von Tresckow J, Koenigsmann M, Gaska T, Kaiser U, Harich HD, Fischer K, Eichhorst B, Hallek M, Fink AM. Second primary malignancies in treated and untreated patients with chronic lymphocytic leukemia. Am J Hematol. 2021 Dec 1;96(12):E457-E460. doi: 10.1002/ajh.26363. Epub 2021 Oct 8. No abstract available. PMID 34591989
- [Derived] von Tresckow J, Heyl N, Robrecht S, Giza A, Aldaoud A, Schlag R, Klausmann M, Linde H, Stein W, Schwarzer A, Fischer K, Cramer P, Eichhorst B, Hallek M, Fink AM. Treatment with idelalisib in patients with chronic lymphocytic leukemia - real world data from the registry of the German CLL Study Group. Ann Hematol. 2023 Nov;102(11):3083-3090. doi: 10.1007/s00277-023-05314-2. Epub 2023 Jun 26. PMID 37358640
- See also: Click here for more information about this study: Registry of the German CLL Study Group — https://www.dcllsg.com/dcllsg-register/